CLINICAL TRIAL: NCT06941415
Title: Bumetanide vs. Furosemide for Adults Hospitalized With Cirrhosis: the BUFF Trial
Brief Title: Bumetanide vs. Furosemide in Cirrhosis
Acronym: BUFF
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stacy Johnson (Other)
Responsible Party: Sponsor-Investigator, Stacy Johnson, Professor of Medicine, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00186841
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Cirrhosis
Keywords: cirrhosis; volume overload; diuresis; furosemide; bumetanide
MeSH Terms: conditions — Fibrosis; Edema | interventions — Bumetanide; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bumetanide (Experimental)
  Interventions: Drug: Bumetanide
- Furosemide (Experimental)
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Bumetanide — Standard of care treatment with bumetanide (intravenous or oral administration) per treating clinician's orders
  Arms: Bumetanide
Drug: Furosemide — Standard of care treatment with furosemide (intravenous or oral administration) per treating clinician's orders
  Arms: Furosemide

SUMMARY:
Patients with cirrhosis are frequently hospitalized due to an acute decompensation of their liver disease including bleeding, jaundice, encephalopathy, and volume overload. Volume overload is associated with increased mortality from acute hypoxic respiratory failure, hemorrhage from esophageal varices, and spontaneous bacterial peritonitis.

Clinical practice guidelines describe sodium restriction and diuretics as first-line treatment, combined with regular body weight monitoring to assess response. In patients with suboptimal response to furosemide, alternative loop diuretics like torsemide or bumetanide may improve natriuresis. Bumetanide has a theoretic advantage over furosemide due to its more rapid and complete intestinal absorption, combined with a prolonged half-life in patients with hepatic dysfunction. In this pragmatic study, the aim is to compare the efficacy of diuresis with bumetanide versus furosemide among hospitalized patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* History of liver cirrhosis
* Clinician placed an order for bumetanide or furosemide in electronic health record within 24 hours of presentation to the hospital

Exclusion Criteria:

* Allergy to bumetanide or furosemide
* Contraindication to diuretic administration (e.g. active bleeding, clinical suspicion of hepatorenal syndrome, hypotension)
* Incarcerated or in custody of law enforcement
* Diuretic ordered for purpose other than volume overload (e.g. hyperkalemia, continuation of home medication without clinical signs of volume overload)
* Inpatient admission not anticipated
* Not admitted to an inpatient hospital bed following initial evaluation in the emergency department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Percent change in weight | 7 days
  Percent change in weight measured in kilograms from date of emergency department presentation (Day 0) to Day 7 of hospitalization, or date of discharge, whichever is earlier

SECONDARY OUTCOMES:
Development of acute kidney injury | 14 days
  Stage 2 or higher acute kidney injury developing within 14 days of presentation to emergency department in accordance with KDIGO criteria
Need for replacement therapy | 14 days
  New initiation of intermittent or continuous hemodialysis within 14 days of presentation to the emergency department
Severe electrolyte derangement | 14 days
  New decrease in serum potassium to less than 2.5 mEq/L within 14 days of presentation to the emergency department
Hospital length of stay | 30 days
  Time from initial presentation to the emergency department to the time of discharge from the hospital or time of death, if a subject dies within the hospital
Unplanned hospital readmission | 30 days
  Readmission to the hospital for an unexpected reason within 30 days of a prior hospital admission
30-day mortality | 30 days
  Death occurring within the 30 days following presentation to the emergency department and subsequent hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Stacy A Johnson, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Findings from the study will be presented at one or more scientific conferences. Results will be submitted for publication to a peer-reviewed journal. Data will be made available to other researchers after publication upon request and local institutional approval.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Following publication of manuscript
Access Criteria: Written request and local institutional approval